CLINICAL TRIAL: NCT04227639
Title: T-piece Versus Pressure-support for the Spontaneous Breathing Trial Before Extubation in Patients at High-risk of Reintubation: a Multicenter Randomized Controlled Trial
Brief Title: T-piece Versus Pressure-support for the Spontaneous Breathing Trial
Acronym: TiP-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TiP-Ex; 2019-A02151-56 (Other: ID-RCB)
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Weaning From Mechanical Ventilation; Extubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-piece trial (Active Comparator): In patients assigned to control group all spontaneous breathing trials will be performed using T-piece trial.
  Interventions: Procedure: T-piece trial
- Pressure-Support trial (Experimental): In patients assigned to experimental group all spontaneous breathing trials will be performed with a pressure-support level of 8 cm H2O without positive end-expiratory pressure.
  Interventions: Procedure: Pressure-support trial

INTERVENTIONS:
Procedure: T-piece trial — T-piece trial will be performed for around 1 hour with a T-piece connected to the extremity of the endotracheal tube by simply disconnecting the patient from the ventilator and by providing additional oxygen (≤ 6 L/min)
  Arms: T-piece trial
Procedure: Pressure-support trial — Pressure-Support trial will be performed for around 1 hour without disconnecting the patient from the ventilator, by using a low level of pressure-support (PS 8 cm H2O) with a FiO2 ≤ 40% and without positive end-expiratory pressure (PEEP), while continuously monitoring the respiratory rate and tidal volume on the ventilator display.
  Arms: Pressure-Support trial

SUMMARY:
The main objective will be to compare the number of ventilator-free days within the 28 days following the first spontaneous breathing trial between strategies of extubation performing spontaneous breathing trials with T-piece trials or with Pressure-Support trials.

To do that, the study director proposed to conduct a prospective multicenter randomized controlled open-label trial comparing these 2 strategies of weaning in patients at high-risk of extubation failure in the Intensive Care Unit.

Patients included will be randomized before performing the first spontaneous breathing trial and will be assigned to one of the following two groups according to the weaning strategy: T-piece trial group or Pressure-Support trial group.

ELIGIBILITY:
Inclusion Criteria:

1. Duration of mechanical ventilation prior to the first spontaneous brathing trial > 24h
2. Patients at high-risk of reintubation according to the following criteria: Patients older than 65 years, or those having any underlying chronic cardiac or lung disease.
3. Patient meeting all weaning criteria according to the international conference consensus on weaning.

   * Respiratory rate ≤ 35 breaths per minute,
   * Adequate oxygenation defined as SpO2 > 90% with FiO2 ≤ 0.4 or PaO2/FiO2 > 150 mm Hg with positive end-expiratory pressure (PEEP) ≤ 8 cmH2O,
   * Adequate cough,
   * Patient awake with a Richmond Agitation-Sedation Scale between +1 and -2
   * No continuous sedation,
   * Hemodynamic stability with no need for vasopressors (or minimal dosis).
4. Informed consent given by the relatives or the patient himself.

Exclusion Criteria:

1. Patients admitted for traumatic brain injury
2. Pre-existing peripheral neuromuscular disease (underlying myopathy or myasthenia gravis)
3. Do-not-reintubate order at time of the first spontaneous breathing trial
4. Patient previously included in the study
5. No Health insurance coverage
6. People under protection: Pregnant or breastfeeding women, minor patients, subjects with guardianship or under law protection.
7. Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days at day 28 | Day 28
  The number of ventilator-free days at day 28, defined as the number of days alive and without invasive mechanical ventilation (intubation or tracheostomy) between the first spontaneous breathing trial (day 1) and day 28.

SECONDARY OUTCOMES:
The number of days alive and without mechanical ventilation (including intubation or non-invasive ventilation) between the first spontaneous breathing trial (day 1) and day 28. | Between Day 1 and Day 28
The number of patients extubated within the 72 hours and within the 7 days following the first spontaneous breathing trial. | Hour 72, Day 7
The number of patients extubated after simple (24h), difficult (> 24 hours and ≤ 7 days) or prolonged ( > 7 days) weaning | Day 28
The number of patients extubated after the first spontaneous breathing trial and not reintubated within the following 72 hours. | Hour 72
The number of days between the first spontaneous breathing trial and the first extubation attempt among extubated patients | Day 28
The number of patients reintubated within the 72 hours and within the 7 days following extubation. | Day 28
The number of patients with post-extubation respiratory failure within the 7 days following extubation. | Day 28
Length of stay in ICU in days. | Day 90
Numbers of patients died in ICU, at day 28 and at day 90. | Day 28 and Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud W. THILLE, Pr, Principal Investigator — CHU Poitiers
Locations (1):
- Intensive reanimation, Poitiers, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available after reasonable request and it has been discussed among the steering committee

REFERENCES:
- [Derived] Metais M, Frat JP, Ehrmann S, Pene F, Decavele M, Terzi N, Prat G, Martin M, Contou D, Gacouin A, Bourenne J, Girault C, Vinsonneau C, Dellamonica J, Labro G, Jochmans S, Herbland A, Quenot JP, Devaquet J, Benzekri D, Ragot S, Thille AW, Coudroy R; FLORALI-IM study group and the REVA Research Network. Factors associated with ICU mortality and long-term outcomes in immunocompromised patients admitted to the intensive care unit for acute respiratory failure. Ann Intensive Care. 2025 Oct 30;15(1):175. doi: 10.1186/s13613-025-01578-1. PMID 41168567
- [Derived] Coudroy R, Lejars A, Rodriguez M, Frat JP, Rault C, Arrive F, Le Pape S, Thille AW. Physiologic Effects of Reconnection to the Ventilator for 1 Hour Following a Successful Spontaneous Breathing Trial. Chest. 2024 Jun;165(6):1406-1414. doi: 10.1016/j.chest.2024.01.038. Epub 2024 Jan 29. PMID 38295948
- [Derived] Thille AW, Gacouin A, Coudroy R, Ehrmann S, Quenot JP, Nay MA, Guitton C, Contou D, Labro G, Reignier J, Pradel G, Beduneau G, Dangers L, Saccheri C, Prat G, Lacave G, Sedillot N, Terzi N, La Combe B, Mira JP, Romen A, Azais MA, Rouze A, Devaquet J, Delbove A, Dres M, Bourenne J, Lautrette A, de Keizer J, Ragot S, Frat JP; REVA Research Network. Spontaneous-Breathing Trials with Pressure-Support Ventilation or a T-Piece. N Engl J Med. 2022 Nov 17;387(20):1843-1854. doi: 10.1056/NEJMoa2209041. Epub 2022 Oct 26. PMID 36286317
- [Derived] Thille AW, Coudroy R, Gacouin A, Ehrmann S, Contou D, Dangers L, Romen A, Guitton C, Lacave G, Quenot JP, Lacombe B, Pradel G, Terzi N, Prat G, Labro G, Reignier J, Beduneau G, Dellamonica J, Nay MA, Rouze A, Delbove A, Sedillot N, Mira JP, Bourenne J, Lautrette A, Argaud L, Levrat Q, Devaquet J, Vivier E, Azais MA, Leroy C, Dres M, Robert R, Ragot S, Frat JP; REVA research network. T-piece versus pressure-support ventilation for spontaneous breathing trials before extubation in patients at high risk of reintubation: protocol for a multicentre, randomised controlled trial (TIP-EX). BMJ Open. 2020 Nov 24;10(11):e042619. doi: 10.1136/bmjopen-2020-042619. PMID 33234658